CLINICAL TRIAL: NCT01264705
Title: A Phase I/II Study of Bavituximab and Sorafenib In Patients With Advanced Hepatocellular Carcinoma
Brief Title: Study of Bavituximab and Sorafenib In Patients With Advanced Liver Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Adam Yopp, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU 062010-150
Record Dates: First submitted 2010-12-01; First posted 2010-12-22 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: Cirrhosis; GI Cancer; Hepatitis; Oncology
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Fibrosis; Gastrointestinal Neoplasms; Hepatitis; Neoplasms | interventions — bavituximab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bavituximab:0.3 mg/kg weekly Sorafenib: 400mg PO twice daily (Experimental): Cohort 1: Participants were administered Bavituximab:0.3 mg/kg weekly Sorafenib: 400mg PO twice daily
  Interventions: Drug: bavituximab (0.3 mg/kg) and sorafenib
- Bavituximab: 1.0 mg/kg weekly Sorafenib: 400mg PO twice daily (Experimental): Cohort 2: Participants were administered Bavituximab:1.0 mg/kg weekly Sorafenib: 400mg PO twice daily
  Interventions: Drug: bavituximab (1.0 mg/kg ) and sorafenib
- Bavituximab: 3.0 mg/kg weekly Sorafenib: 400mg PO twice daily (Experimental): Cohort 3: Participants were administered Bavituximab:3.0 mg/kg weekly Sorafenib: 400mg PO twice daily
  Interventions: Drug: bavituximab (3.0 mg/kg) and sorafenib

INTERVENTIONS:
Drug: bavituximab (0.3 mg/kg) and sorafenib — Bavituximab:0.3 mg/kg weekly Sorafenib: 400mg PO twice daily
  Arms: Bavituximab:0.3 mg/kg weekly Sorafenib: 400mg PO twice daily
Drug: bavituximab (1.0 mg/kg ) and sorafenib — Bavituximab: 1.0 mg/kg weekly Sorafenib: 400mg PO twice daily
  Arms: Bavituximab: 1.0 mg/kg weekly Sorafenib: 400mg PO twice daily
Drug: bavituximab (3.0 mg/kg) and sorafenib — Bavituximab: 3.0 mg/kg weekly Sorafenib: 400mg PO twice daily
  Arms: Bavituximab: 3.0 mg/kg weekly Sorafenib: 400mg PO twice daily

SUMMARY:
This is a non-randomized, open-label, single-institution phase I/II therapeutic trial of bavituximab and sorafenib in patients with advanced hepatocellular carcinoma (HCC). This study will be activated at the UT Southwestern Medical Center, comprised of The Harold C. Simmons Comprehensive Cancer Center, UT Southwestern Hospitals-St. Paul and Parkland Memorial Hospital System. Advanced HCC is defined as disease that is not amenable to surgical resection or orthotopic liver transplantation or is metastatic in nature.

DETAILED DESCRIPTION:
The investigators are looking for men or women aged 18 years or older with hepatocellular carcinoma not suitable for surgical resection or hepatic transplantation. Prior locoregional therapy including but not limited to transarterial chemoembolization (TACE), radiofrequency ablation (RFA) or ethanol injection is allowed as long as the treatment was 4 weeks previous. Patients must be Child-Pugh A with no previous treatment with sorafenib or other vascular endothelial growth factor (VEGF) inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of hepatocellular carcinoma by at least one criterion listed below:

   * Histologically confirmed.
   * MRI or CT consistent with liver cirrhosis and at least one solid liver lesion >2 cm with early enhancement and delayed enhancement washout regardless of AFP.
   * AFP >400 ng/ml and evidence of at least one solid liver lesion >2 cm regardless of specific imaging characteristics on CT or MRI.
2. Locally advanced or metastatic disease.
3. Patients with locally advanced disease must have disease deemed to be unresectable or not eligible for hepatic transplantation. Determination will occur in the weekly GI DMT meeting by surgical oncologists and transplant surgeons.
4. Measurable disease, as defined as lesions that can accurately be measured in at least one dimension (longest diameter to be measured) according to Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1) at least 2 cm with conventional techniques or at least 1 cm with spiral computed tomography.
5. Child-Pugh Score A.
6. Age ≥ 18 years.
7. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-2.
8. Absolute neutrophil count ≥ 1,500 cells/mm3.
9. Platelet count ≥ 75,000 cells/mm3.
10. Total bilirubin ≤ 3.0 mg/dl.
11. Hemoglobin ≥ 8.5 g/dl.
12. AST and ALT ≤ 5.0 times upper limit of normal.
13. D-dimer ≤ 3 times upper limit of normal.
14. INR ≤ 1.8 (therapeutic anticoagulation allowed as long as medically indicated.

Exclusion Criteria:

1. History of bleeding diathesis or coagulopathy.
2. Symptomatic or clinically active brain metastases.
3. Major surgery within previous 4 weeks.
4. History of thromboembolic events (including both pulmonary embolisms and deep vein thrombosis); central venous catheter-related thrombosis > 6 months prior is allowed.
5. Prior adjuvant therapy with sorafenib or other Raf/MEK/RAS or VEGFR inhibitors. Prior adjuvant therapy is allowed provided it was completed > 6 months ago and there is documented recurrence of hepatocellular carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-01; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam C Yopp, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Mokdad AA, Zhu H, Beg MS, Arriaga Y, Dowell JE, Singal AG, Yopp AC. Efficacy and Safety of Bavituximab in Combination with Sorafenib in Advanced Hepatocellular Carcinoma: A Single-Arm, Open-Label, Phase II Clinical Trial. Target Oncol. 2019 Oct;14(5):541-550. doi: 10.1007/s11523-019-00663-3. PMID 31429027

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bavituximab:0.3 mg/kg Weekly Sorafenib: 400mg PO Twice Daily | Bavituximab: 1.0 mg/kg Weekly Sorafenib: 400mg PO Twice Daily | Bavituximab: 3.0 mg/kg Weekly Sorafenib: 400mg PO Twice Daily
Started | 3 | 3 | 41
Completed | 3 | 3 | 41
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bavituximab:0.3 mg/kg Weekly Sorafenib: 400mg PO Twice Daily | Bavituximab: 1.0 mg/kg Weekly Sorafenib: 400mg PO Twice Daily | Bavituximab: 3.0 mg/kg Weekly Sorafenib: 400mg PO Twice Daily | Total
Number analyzed (Participants) | 3 | 3 | 41 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 33 | 37
  >=65 years | 1 | 1 | 8 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 7 | 9
  Male | 2 | 2 | 34 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1 | 0 | 16 | 17
  White | 1 | 0 | 13 | 14
  Hispanic | 1 | 2 | 10 | 13
  Asian | 0 | 1 | 2 | 3
  Unknown | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Median Radiographic Time to Progression (TTP) Calculated From Treatment Initiation to First Evidence of Disease Progression or Last Follow-up.
Description: Median radiographic time to progression (TTP) was calculated from treatment initiation to first evidence of disease progression or last follow-up by using the Kaplan-Meier method. The 95% confidence intervals (CIs) for time-to-progression data was calculated using Greenwood's formula.
Time Frame: Treatment initiation to first evidence of disease progression or last follow-up, an average of 24 months
Population: Cohort 1 and 2 were part of phase 1 study and at the phase 1 study this outcome was not collected. The 3 participants who received dose Bavituximab: 3.0 mg/kg weekly Sorafenib: 400mg PO twice daily were part of phase 1 and hence they were not part of phase 2 . Hence their data were not analyzed here.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cohort 1: Bavituximab:0.3 mg/kg weekly Sorafenib: 400mg PO twice daily
- Cohort 2: Bavituximab: 1.0 mg/kg weekly Sorafenib: 400mg PO twice daily
- Cohort 3: Bavituximab: 3.0 mg/kg weekly Sorafenib: 400mg PO twice daily
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 38
months |  |  | 6.7 [4.1 to 16.9]

2. Primary Outcome: Number of Patients With Dose Limiting Toxicity
Description: Dose limiting toxicity by serious adverse events by CTCAE version 4.0
Time Frame: 8 months.
Population: This outcome was for phase 1 only
Measure: Number; unit: participants
Arm/Group | Bavituximab:0.3 mg/kg Weekly Sorafenib: 400mg PO Twice Daily | Bavituximab: 1.0 mg/kg Weekly Sorafenib: 400mg PO Twice Daily | Bavituximab: 3.0 mg/kg Weekly Sorafenib: 400mg PO Twice Daily
Number analyzed (Participants) | 3 | 3 | 3
participants | 0 | 0 | 0

3. Secondary Outcome: Safety, as Measured by the Number of Patients With Adverse Event Related to the Treatment That Experienced Grade 3 or Greater.
Description: Safety was measured by the number of patients with at least one adverse event as assess by NCI Common Terminology criteria for adverse events (CTCAE)
Time Frame: Up to 3 months of patient enrollment (phase 1)
Population: This outcome measure was only analyzed for phase 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

4. Secondary Outcome: Median Months of Overall Survival Calculated From Treatment Initiation to Death or Last Follow-up.
Description: Median months of overall survival was calculated from treatment initiation to death or last follow-up by using the Kaplan-Meier method. The 95% confidence intervals (CIs) for median months of overall survival was calculated using Greenwood's formula.
Time Frame: Treatment initiation to death or last follow-up, an average 24 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 38
months |  |  | 6.1 [4.9 to 8.1]

5. Secondary Outcome: Median Months of Disease Specific Survival Calculated From Treatment Initiation to Death From Advanced HCC (Hepatocellular Carcinoma) or Last Follow-up.
Description: Median months of disease specific survival was calculated from treatment initiation to first evidence of death from advanced liver cancer or last follow-up by using the Kaplan-Meier method. The 95% confidence intervals (CIs) for time-to-disease specific survival data was calculated using Greenwood's formula.
Time Frame: Treatment initiation to first evidence of death from advanced liver cancer or last follow-up, an average of 12 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 38
months |  |  | 8.6 [6.2 to 13.5]

ADVERSE EVENTS:
Time Frame: SAEs and Other AEs were monitored up to 8 months (Phase 1) SAEs and Other AEs were monitored up to 2 years (Phase 2)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 38/41
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/41
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 12/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=41)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 12 (12)
fatigue (General disorders) | 0 (0) | 0 (0) | 10 (10)
anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 9 (9)
abdominal cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (7)
hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 5 (5)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Hand /foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
nausea (General disorders) | 0 (0) | 0 (0) | 3 (3)
Gerd (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
stomstitis (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
infusion reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
hiccoughs (General disorders) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT01264705/Prot_SAP_000.pdf